CLINICAL TRIAL: NCT03330821
Title: Phase 1B/II Study of Escalating Doses of Pevonedistat (TAK-924, Formerly MLN4924) Administered in Combination With Standard Induction Chemotherapy (Cytarabine and Idarubicin) in Newly Diagnosed High Risk Acute Myelogenous Leukemia (AML)
Brief Title: Pevonedistat, Cytarabine, and Idarubicin in Treating Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-17-6; NCI-2017-01710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-17-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: interventions — Cytarabine; Idarubicin; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (idarubicin, cytarabine, pevonedistat) (Experimental): INDUCTION: Patients receive idarubicin IV over 10-15 minutes on days 1-3, cytarabine IV over 1-3 hours on days 1-7, and pevonedistat IV over 60 minutes on days 1, 3, and 5. Patients with gross residual disease on day 14 bone marrow may receive a second course of induction chemotherapy.
  CONSOLIDATION: Patients who achieve CR and will not undergo bone marrow transplant receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats every 28-35 days for 4 courses in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Other: Laboratory Biomarker Analysis; Drug: Pevonedistat; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of pevonedistat and to see how well it works in combination with cytarabine and idarubicin in treating patients with acute myeloid leukemia. Pevonedistat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Given pevonedistat, cytarabine, and idarubicin may work better in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of pevonedistat in combination with cytarabine and idarubicin in newly diagnosed high-risk acute myeloid leukemia. (Phase Ib) II. To determine the composite complete response rate (complete remission [CR] or complete remission with incomplete blood count recovery [CRi]) of pevonedistat in combination with cytarabine and idarubicin in newly diagnosed high-risk acute myeloid leukemia. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate plasma pharmacokinetic (PK) profiles of pevonedistat when used in combination with cytarabine and idarubicin in the phase Ib part of the study.

II. To evaluate the relapse free (RFS), overall survival (OS), safety and tolerability of pevonedistat in combination with cytarabine and idarubicin in the phase II part of the study.

TERTIARY OBJECTIVES:

I. To evaluate the pharmacodynamics (PD) effects of pevonedistat in combination with cytarabine and idarubicin in acute myelogenous leukemia (AML) blasts.

II. To evaluate potential predictive biomarkers of response to pevonedistat in combination with cytarabine and idarubicin in AML.

III. To determine the CR without minimal residual disease rate (CR MRD-) of pevonedistat in combination with cytarabine and idarubicin in newly diagnosed acute myeloid leukemia.

OUTLINE: This is a phase Ib, dose escalation study of pevonedistat followed by a phase II study.

INDUCTION: Patients receive idarubicin intravenously (IV) over 10-15 minutes on days 1-3, cytarabine IV over 1-3 hours on days 1-7, and pevonedistat IV over 60 minutes on days 1, 3, and 5. Patients with gross residual disease on day 14 bone marrow may receive a second course of induction chemotherapy.

CONSOLIDATION: Patients who achieve CR and will not undergo bone marrow transplant receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats every 28-35 days for 4 courses in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up for at least 30 days, and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 1 highly effective method and 1 additional (barrier) of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only and lactational amenorrhea are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (ie, status postvasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), or
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only and lactational amenorrhea are not acceptable methods of contraception)
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0-2
* Expected survival > 3 months from study enrollment
* Within 3 days before the first dose of study drug: albumin > 2.7 g/dL
* Within 3 days before the first dose of study drug: total bilirubin < upper limit of normal (ULN)
* Within 3 days before the first dose of study drug: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN
* Within 3 days before the first dose of study drug: creatinine clearance > 50 mL/min
* Within 3 days before the first dose of study drug: hemoglobin > 8 g/dL (prior red blood cell [RBC] transfusion allowed); patients may be transfused to achieve this value; elevated indirect bilirubin due to post-transfusion hemolysis is allowed
* Patients with previously untreated AML (except acute promyelocytic leukemia [APL]) who have at least one of the following:

  * Adverse genetic features as per the European Leukemia Net guidelines
  * Treatment related AML or AML with antecedent myelodysplastic syndrome (MDS); (patient who have received treatment with hypomethylating agents for MDS and have now transformed to AML are eligible)
  * Are over the age of 55 years and considered fit for chemotherapy
  * Patients with AML with MDS-related changes
* Patients must be considered candidates for intensive chemotherapy treatment with standard doses of cytarabine and anthracycline regimen (?7+3 regimen?)
* White blood cell (WBC) count < 50,000/uL before administration of pevonedistat on cycle 1 day 1; Note: hydroxyurea may be used to control the level of circulating leukemic blast cell counts to not lower than 10,000/uL during the study

Exclusion Criteria:

* Known cardiopulmonary disease defined as one of the following:

  * Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)
  * Cardiomyopathy or history of ischemic heart disease
  * Arrhythmia (eg, history of polymorphic ventricular fibrillation or torsade de pointes); however, patients with < grade 3 atrial fibrillation (a fib) for a period of at least 6 months may enroll; grade 3 a fib is symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation; patients with paroxysmal a fib are permitted to enroll
  * Implantable cardioverter defibrillator
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV; or class II with a recent decompensation requiring hospitalization or referral to a heart failure clinic within 4 weeks before screening), myocardial infarction and/or revascularization (eg, coronary artery bypass graft, stent) within 6 months of first dose of study drug
  * Patients who had ischemic heart disease who have had acute coronary syndrome (ACS), myocardial infarction (MI), and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll
  * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing)
  * Pulmonary hypertension
* Prolonged rate corrected QT (QTc) interval >= 500 msec, calculated according to institutional guidelines
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography
* Known moderate to severe chronic obstructive pulmonary disease (COPD), interstitial lung disease, and pulmonary fibrosis
* Any serious medical or psychiatric illness that could, in the investigator?s opinion, potentially interfere with the completion of study procedures
* Treatment with any investigational products within 14 days before the first dose of any study drug
* Patients receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy within 14 days of first receipt of study drug with the exception of: hydroxyurea (HU) in patients who need to continue this agent to maintain WBC count =< 50,000/mm^3
* Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, septicemia, or methicillin resistant staphylococcus aureus infection
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period
* Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection
* Life-threatening illness unrelated to cancer
* Patients with uncontrolled coagulopathy or bleeding disorder
* Known central nervous system (CNS) involvement
* Known human immunodeficiency virus (HIV) seropositive
* Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection

  * Note: patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load
* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Systemic antineoplastic therapy or radiotherapy within 14 days before the first dose of any study drug, except for hydroxyurea
* Treatment with clinically significant metabolic enzyme inducers within 14 days before the first dose of the study drug; clinically significant metabolic enzyme inducers are not permitted during this study
* Patients who refuse to potentially receive blood products and/or have a hypersensitivity to blood products
* Patients with history of allergic or toxic reactions attributed to cytarabine or a history of allergic reactions to components of the formulated product
* Patients with history of allergic or toxic reactions attributed to anthracyclines or a history of allergic reactions to components of the formulated product
* Patients who have had prior chemotherapy for AML
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s)
* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on day 1 before first dose of study drug (if applicable)
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite complete response rate | Up to 2 years
  Response will be assessed according to the 2017 European Leukemia Net Guidelines. The composite complete response rate will be calculated as the percentage of patients who have CR or CRi. Wilson 95% confidence interval will be provided.
Incidence of adverse events (Phase Ib) | Up to 22 days
  Will be assessed by Common Terminology Criteria for Adverse Events version 4.03.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | From the date of achievement of a remission until the date of relapse or death from any cause, assessed up to 2 years
  RFS will be calculated as the date of achievement of a remission (CR or CRi) until the date of relapse (documented morphological recurrence (≥ 5% blasts on in the bone marrow, reappearance of blasts in the blood or development of extramedullary disease after CR) or death - whichever comes first; patients who are alive and have not progressed or recurred at the time of their last disease assessment, will be censored at that time. Survival curves will be plotted by the Kaplan-Meier (KM) method. Median RFS and their 95% confidence intervals, 1-year and 2- year survival rates and corresponding standard errors will be derived from the KM curves.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kelly, MD, Principal Investigator — University of Southern California
Locations (5):
- United States (5):
  - University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Cleveland Clinic, Cleveland, Ohio